CLINICAL TRIAL: NCT02668887
Title: A Prospective Cohort Study on Employment and Quality of Life in Patients With Malignant Melanoma
Brief Title: Employment and Quality of Life in Patients With Malignant Melanoma
Status: Completed | Type: Observational
Sponsor: Fachklinik Hornheide an der Universität Münster (Other)
Collaborators: Universität Münster (Other); Deutsche Rentenversicherung (Other)
Responsible Party: Principal Investigator, Susanne Dugas-Breit, M.D., Fachklinik Hornheide an der Universität Münster
Other Study IDs: Hornheide-Derm-001
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Malignant Melanoma of Skin; Quality of Life; Work Ability
MeSH Terms: conditions — Melanoma | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Quality of Life, status of employment

SUMMARY:
Within the first year after diagnosis, data on employment and quality of life will be collected and evaluated in patients with malignant melanoma

ELIGIBILITY:
Inclusion Criteria:

* first diagnosis of malignant melanoma stage 0 to stage IIIC within the last 6 weeks
* written informed consent

Exclusion Criteria:

* diagnosis of malignant melanoma stage IV
* inability to follow the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant melanoma
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joachim Schulze, M.D., Study Director — Fachklinik Hornheide
Locations (1):
- Fachklinik Hornheide, Münster, Germany

IPD SHARING:
Plan to Share IPD: No